CLINICAL TRIAL: NCT04130516
Title: A Multicenter Phase 1-2A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of LNS8801 in Patients With Advanced Cancer With and Without Pembrolizumab
Brief Title: Study Assessing MTD, Safety, Tolerability, PK and Anti-tumor Effects of LNS8801alone and With Pembrolizumab
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Linnaeus Therapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNS-101; MK3475-B47 (Other: Merck, Sharpe and Dohme, LLC); KEYNOTE-B47 (Other: Merck, Sharpe and Dohme, LLC)
Record Dates: First submitted 2019-10-10; First posted 2019-10-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult
Keywords: Melanoma, Uveal Melanoma, NSCLC, Colorectal, Pancreatic, and Gastric Cancers
MeSH Terms: conditions — Melanoma; Uveal Melanoma; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Other): Phase 1/2 open-label
  Interventions: Drug: LNS8801 -Small molecule, orally bioavailable, selective agonist of GPER; Biological: Pembrolizumab - anti-PD-1 antibody

INTERVENTIONS:
Drug: LNS8801 -Small molecule, orally bioavailable, selective agonist of GPER — LNS8801 -Small molecule, orally bioavailable, selective agonist of GPER
Biological: Pembrolizumab - anti-PD-1 antibody — pembrolizumab- anti-PD-1 antibody
  Other Names: KEYTRUDA®; Pembrolizumab

SUMMARY:
This Phase 1/2, first-in-human, open-label, multicenter study follows a 3+3 ascending dose escalation design to determine the MTD/RP2D and to characterize the safety, tolerability, PK, and antitumor effects of LNS8801 alone and in combination with pembrolizumab. The study will include a dose escalation phase, a dose expansion phase, and phase 2A cohorts. Up to 200 patients will be accrued for this study. Up to 15 study sites in the United States will participate in the study.

DETAILED DESCRIPTION:
In this Phase 1/2, first-in-human, open-label, multi-center study. Dose escalation cohorts enrolled at least 3 patients in accordance with a traditional dose escalation 3+3 design, and the study will determine the MTD/RP2D of LNS8801. LNS8801 will be administered orally 3 days/week or once or twice a day during 21 day cycles until disease progression or unacceptable toxicity occurs.

Safety assessments will be performed on all patients at screening, throughout their participation in the study, and for 30 days (90 days in combination cohorts) following the last dose of study drug. Throughout the study, imaging of tumors for evidence of tumor response and/or progression will be performed; biopsies will be performed on accessible lesions.

After the RP2D of LNS8801 is identified and the safety of dosing LNS8801 with pembrolizumab has been established, expansion cohorts and Phase 2A cohorts will open. Any 2 dose escalation cohorts may be expanded to 8 to 10 patients to include additional patients to further explore PK and PD.

Phase 1B expansion cohorts include a monotherapy cohort (LNS8801 alone) of melanoma patients (not uveal) who are now not eligible for additional anti-PD-1 therapy in the judgement of the investigator because of prior severe immune related adverse events and a combination therapy (LNS8801 + pembrolizumab) cohort in anti-PD-1/L1 refractory advanced cancer patients who have previously had clinical benefit on anti-PD-1/L1 therapy alone or in combination (complete response or partial response of any duration, or confirmed stable disease for at least 16 weeks) but have since relapsed and not had an intervening cytotoxic chemotherapy. Up to 28 evaluable patients may be studied in each cohort.

The study will also include the following 8 Phase 2A cohorts.

Monotherapy with 125 mg LNS8801 PO:

COHORT M2: up to 20 evaluable patients with no remaining SOC therapies with pancreatic, gastric, non small cell lung cancer (NSCLC) or colorectal cancers.

COHORT M3: up to 10 evaluable patients with no remaining SOC therapies with advanced malignant cutaneous melanoma having received as their immediate prior line of therapy a PD-1/L1 targeted immune checkpoint inhibitor (IO), alone or in combination, and who are now not eligible for anti-PD-1 treatment in the judgement of the Investigator due to prior severe immune related adverse events.

COHORT M4: up to 10 patients with advanced solid tumor malignancies and no remaining SOC therapies, other than cutaneous melanoma, having received as their immediate prior line of therapy a PD-1/L1 targeted immune checkpoint inhibitor (IO), alone or in combination, and having been forced to discontinue IO therapy due to an immune-related adverse event (irAE).

COHORT M5: up to 10 evaluable patients with metastatic uveal melanoma and no remaining SOC therapies that have 2 or fewer prior lines of systemic therapy.

Combination therapy cohorts treated with 125 mg LNS8801 daily PO + 200 mg Q3W Pembrolizumab IV:

COHORT C2: up to 20 evaluable patients with no remaining SOC therapies with pancreatic, gastric, non small cell lung cancer (NSCLC) or colorectal cancers.

COHORT C3: up to 10 evaluable patients with metastatic non-small cell lung cancer (NSCLC) expressing PD-L1 (Tumor Proportion Score [TPS] ≥1% and ≤49%) as determined by an FDA-approved test will be treated with the combination of LNS8801 plus pembrolizumab. Eligible patients must either have no EGFR or ALK genomic tumor aberrations or have not demonstrated disease response on or following FDA-approved therapy for these aberrations. Inclusion and exclusion criteria will otherwise be consistent with those criteria specified above.

COHORT C5: up to 10 evaluable patients with metastatic uveal melanoma and no remaining SOC therapies that have 2 or fewer prior lines of systemic therapy.

COHORT C6: up to 10 evaluable patients with advanced malignant cutaneous melanoma and no remaining SOC therapies.

Up to 200 patients will be accrued for this study at up to 15 study sites in the United States.

ELIGIBILITY:
Prescreening Inclusion Criteria for genotyping:

1. Has histopathologically confirmed locally advanced or metastatic solid tumor cancer.
2. Is able to understand and voluntarily sign a written informed consent form and is willing and able to comply with protocol requirements.
3. Is considered likely to meet the detailed inclusion and exclusion criteria for treatment when required.

Inclusion Criteria for treatment portion of study:

1. Has histopathologically confirmed locally advanced or metastatic solid tumor cancer (or lymphoma in Phase 1). The solid tumor cancer is further defined in some cohorts as:

   1. Phase 1B monotherapy expansion cohort:

      Has melanoma, except uveal melanoma, and has previously received anti-PD-1/L1 therapy and is now not eligible for anti-PD-1 treatment in the judgement of the Investigator due to prior severe immune related adverse events, and has not received intervening cancer therapy since the anti-PD-1/L1 therapy.
   2. Monotherapy Cohort M2:

      Has pancreatic, gastric, non small cell lung cancer (NSCLC), or colorectal cancer.
   3. Monotherapy Cohort M3:

      Has cutaneous melanoma, and has previously received anti-PD-1/L1 therapy and is now not eligible for anti-PD-1 treatment in the judgement of the Investigator due to prior severe immune related adverse events, and has not received intervening cancer therapy since the anti-PD-1/L1 therapy.
   4. Monotherapy Cohort M4:

      Has any solid tumor malignancy, except cutaneous melanoma, and has previously received anti-PD-1/L1 therapy and is now not eligible for anti-PD-1 treatment in the judgement of the Investigator due to prior severe immune related adverse events, and has not received intervening cancer therapy since the anti-PD-1/L1 therapy.
   5. Monotherapy Cohort M5:

      Has metastatic uveal melanoma, and has received ≤ 2 prior lines of prior systemic therapy.
   6. Phase 1B combination expansion cohort:

      Has any locally advanced or metastatic solid tumor cancer, and has first had a clinical benefit from, followed by documented disease progression on an anti-PD-1/L1 treatment administered either as monotherapy or in combination. Clinical benefit is defined as a complete or partial response of any duration or stable disease for at least 16 weeks with at least one scan showing stable disease. Patients should not have received intervening therapy that did not include anti-PD1/L1 between finishing anti-PD-1/L1 treatment and commencing study treatment.

      Disease progression on an anti-PD-1/L1 therapy is defined as both:
      1. Having received anti-PD-1/L1 therapy at least twice if dosed every 4 weeks (q4w) or longer, at least 3 times if dosed every 3 weeks (q3w), or at least 4 times if dosed every 2 weeks (q2w) and,
      2. Having documented clinical or radiographic progression of disease (PD) while on anti-PD-1/L1 therapy.
   7. Combination Therapy Cohort C2:

      Has pancreatic, gastric, NSCLC, or colorectal cancer.
   8. Combination Therapy Cohort C3:

      Has metastatic NSCLC expressing PD-L1 with a Tumor Proportion Score (TPS) ≥1% and ≤49% as determined by an FDA-approved test, and must not have EGFR or ALK genomic tumor aberrations or have demonstrated disease response on or following FDA-approved therapy for these aberrations, and is PD-1/L1 naïve, and is eligible for pembrolizumab as the standard of care or has no available standard of care.
   9. Combination Therapy Cohort C5:

      Has metastatic uveal melanoma and, has received ≤ 2 prior lines of prior systemic therapy.
   10. Combination Therapy Cohort C6:

   Has cutaneous melanoma.
2. Has no standard of care or the patient declines standard of care options.

   a. An exception to this is metastatic NSCLC patients expressing PD-L1 with a Tumor Proportion Score (TPS) ≥1% and ≤49% who may enter Phase 2 pembrolizumab Combination Therapy Cohort C3 with anti-PD-1 therapy as their standard of care.
3. Has measurable disease per RECIST v1.1 or RANO as assessed by the local site investigator/radiologist. Lesions in a previously irradiated area are measurable if progression has been demonstrated after radiation. Lesions must be measurable in at least 2 dimensions in a spiral CT scan or MRI. For lymphoma patients only, the minimum measurement must be >15 mm on the long axis and >10 mm on the short axis.

   a. Patients with RECIST target lesions in bones must have a PET scan between their last cancer therapy and Cycle 1 Day 1.
4. Be at least18 years of age on day of signing informed consent.
5. Have an Eastern Cooperative Oncology Group Performance Status of 0 or 1.
6. Have an estimated life expectancy of >3 months.
7. Patients who have surgically accessible lesions should agree to biopsies from nonirradiated tumor lesions or irradiated tumor lesions that have shown progression since irradiation. For the avoidance of doubt, if no surgically accessible lesions exist or a biopsy is contraindicated, patients may still enter the study.
8. Be able to swallow capsules and tablets.
9. Have adequate organ and bone marrow function defined by:

   1. Absolute neutrophil count >=1.5 × 109/L (>=1500/mm3).
   2. Hemoglobin >=9.0 g/dL or equivalent. Criteria must be met without packed red blood cell transfusion within the prior 2 weeks. Participants can be on a stable dose of erythropoietin (≥ 3 months).
   3. Platelet count >=75 × 10e9/L (>=75,000/mm3) for LNS8801 monotherapy cohorts Platelet count >=100 × 10e9/L (>=100,000/mm3) for LNS8801/pembrolizumab combination cohorts.
   4. Total bilirubin <=1.5 × institutional upper limit of normal (ULN), unless known Gilbert syndrome has been diagnosed.
   5. Measured or calculated creatinine clearance (glomerular filtration rate) >=50 mL/min/1.73 m2.
   6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=2.5 × ULN or <=5 × ULN with cancer in the liver.
   7. For cohorts receiving LNS8801/pembrolizumab combination therapy, prothrombin time (PT) or activated partial thromboplastin time (aPTT) must be ≤1.5 × ULN. If a participant is receiving anticoagulant therapy, PT or aPTT must be within therapeutic range of intended use of anticoagulants.
10. Female patients of childbearing potential must have a negative serum pregnancy test at screening and a negative (serum or urine) pregnancy test within 72 hours before the first dose of study drug. If the urine test is positive or cannot be confirmed negative, a serum pregnancy test will be required and must be negative for the patient to be eligible.
11. Female patients must not be breastfeeding.
12. Female patients of childbearing potential must be willing to use a highly effective contraception method prior to study entry, while on study drug, and for a period of at least 4 months following the last dose of study drug.

    Note: Women receiving estrogen-based contraceptives will be excluded from the study.

    Note: A woman is considered of childbearing potential unless she is postmenopausal (>1 year without menses and confirmed with a follicle-stimulating hormone test) or surgically sterilized via bilateral oophorectomy, hysterectomy, bilateral tubal ligation, or successful Essure® placement with a documented confirmation test at least 3 months after the procedure.

    Male patients must be surgically sterile or willing to use a highly effective double-barrier contraception method (eg, male condom with diaphragm or male condom with cervical cap) upon study entry, while on study drug, and for a period of at least 4 months following the last dose of study drug. Males must agree to refrain from donating sperm during this period.
13. Highly effective contraception is defined as a method of contraception that has a <1% failure rate when used consistently and correctly (as defined by the International Council for Harmonization Guidance on Nonclinical Safety Studies for the Conduct of Human Clinical Research M3 [R2]). These methods include implants, injectables, combined hormonal contraceptives (eg, combined oral contraceptives [excluding estrogen-based contraceptives], patch, and vaginal ring), some intrauterine devices (IUDs) (eg, IUD or intrauterine system), sexual abstinence, or a monogamous relationship with a vasectomized partner.

    a. True abstinence, when in line with the preferred and usual lifestyle of the patient, is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug (ie, 60 days after discontinuing study drug or 5 times the terminal elimination half-life, whichever is longer). Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
14. Be able to understand and voluntarily sign a written informed consent form and is willing and able to comply with protocol requirements.

Exclusion Criteria for Treatment Portion of Study:

1. Has thyroid cancer or gall bladder cancer (excluded from Phase 1 cohorts only).
2. Has any cancer that is known to be estrogen receptor-positive (ERalpha+).
3. Received an anticancer therapy within 4 weeks (6 weeks for nitrosoureas, mitomycin C, or pembrolizumab given on a 6-week cycle) or 5 half-lives, whichever is shorter, before the first dose of study drug. Except in anti-PD-1/L1 refractory cohorts, where patients may start LNS8801 therapy at what would be the beginning of the next cycle of their immunotherapy cycle (eg, LNS8801 may be dosed 3 or 6 weeks after the last dose of pembrolizumab depending on cycle, or 4 weeks after nivolumab) if that is shorter.
4. Has unresolved toxicities from previous anticancer therapy. Anticancer therapy toxicities are defined as toxicities (other than alopecia) not yet resolved according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 ≤ Grade 1, or baseline (participants with ≤ Grade 2 neuropathy may be eligible).

   * Note: Patients in an LNS8801/pembrolizumab combination cohort must not have undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Participants who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of acute graft versus host disease [GVHD])
5. Patients must not be participating in another study of an investigational agent or have used an investigational device within 4 weeks before the first dose of study drug.

   Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
6. Has a symptomatic primary central nervous system (CNS) tumor, symptomatic CNS metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression.

   Note: Patients are eligible if neurologic symptoms and CNS imaging are stable and steroid dose is stable for 14 days prior to the first dose of study drug and no CNS surgery or radiation has been performed for 28 days (14 days if stereotactic radiosurgery).

   a. In a LNS8801/pembrolizumab combination cohorts, has known active CNS metastases and/or carcinomatous meningitis.
7. Requires the use of antitumor necrosis factor (anti-TNF) therapies, such as infliximab, or has received treatment with anti-TNF therapies within 5 half-lives of that therapy.
8. Has an active autoimmune disease that required systemic treatment in the past 2 years (ie, with use of disease-modifying antirheumatic agents or immunosuppressive drugs).

   Note: Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal, thyroid, or pituitary insufficiency) is permitted.
9. Has a diagnosis of immunodeficiency, is on immunosuppressive therapy, or is receiving chronic systemic or enteric steroid therapy (in dosing exceeding 10 mg/day of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

   Note: At screening, patients may be using systemic corticosteroids (dose 10 mg/day of prednisone or equivalent) or topical or inhaled corticosteroids.
10. Is receiving any other investigational agent(s) or has received an investigational agent within 30 days or 5 half-lives, whichever is shorter, of the first dose of study drug.
11. Has had major surgery (excluding placement of vascular access) within 4 weeks prior to the planned start of LNS8801.
12. Has had radiotherapy with a limited field for palliation (less than 2 weeks) within 1 week of the first dose of study drug to non-CNS disease, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation, which must be completed at least 4 weeks prior to the first dose of study drug. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
13. Has evidence of pneumonitis or interstitial lung disease.

    a. For pembrolizumab combination cohorts, has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
14. Has any of the following known infections:

    1. Human immunodeficiency virus (HIV), hepatitis B virus (HBV) (ie, hepatitis B surface antigen-positive), or hepatitis C virus (HCV) (ie, detectable HCV ribonucleic acid [RNA]).

       Note: Patients with a prior history of treated HBV infection who are antigen-negative or patients with a prior history of treated HCV infection who are HCV RNA-undetectable may be enrolled.
    2. Active infections requiring systemic therapy (including asymptomatic infections with positive virus titers and the Investigator's judgment that worsening of the condition is likely with study drug or the condition would impair or prohibit a patient's participation in the study).
15. Has active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug.
16. Has received a live vaccine within 30 days of the planned start of study drug.
17. Has a corrected QT interval (QTc) by Fridericia method >450 msec for male patients or >470 msec for female patients, or a history or risk factors for or use of medications known to prolong the QTc or that may be associated with torsades de pointes.

    Note: Isolated right bundle branch block and incomplete right bundle branch block and left anterior hemiblock are acceptable.
18. Has had any prior treatment for the present solid malignancy with GPER agonists (eg, tamoxifen, raloxifene, or estrogen hormone replacement therapy). History of oral contraceptive use is permissible.
19. Is using a strong inhibitor or inducer of cytochrome P450 1A2, 2C9, 2C19, 2D6, or 3A4.
20. Requires treatment with a proton pump inhibitor.
21. Has received estrogen treatment since cancer diagnosis or the presumed initiation of their cancer, including estrogen-based contraceptives.
22. Has a cancer that was treated with estrogen hormone therapy.
23. Is currently using estrogen hormone replacement therapy, was diagnosed while on estrogen hormone replacement therapy, or has used estrogen replacement therapy since diagnosis.
24. Is pregnant, lactating, has been pregnant within the last 2 years, or is planning to attempt to become pregnant or impregnate someone during this study or within 90 days after dosing of study drug (120 days for LNS8801/pembrolizumab combination cohorts).
25. Has a history of another active malignancy (a second cancer) within the previous 2 years except for localized cancers that are not related to the current cancer being treated, are considered cured, and, in the opinion of the Investigator, presents a low risk of recurrence. These exceptions include, but are not limited to, basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
26. Has an uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, hypertension, unstable angina pectoris, cardiac arrhythmia, autoimmune or inflammatory diseases, or psychiatric illness/social situations that would limit compliance with study requirements.
27. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
28. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study in the medical judgement of the investigator.
29. Has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of trial treatment for patients with non-small cell lung cancer.
30. In the LNS8801/pembrolizumab combination cohorts, has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher irAE.
31. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Adverse events observed for LNS8801 dosed alone and in combination with pembrolizumab | Duration of study, approximately 24 months

SECONDARY OUTCOMES:
LNS8801 plasma exposure (AUC) as a function of dose | During first 23 days of dosing
  AUC0-end
LNS8801 plasma exposure (Cmax) as a function of dose | During the first 23 days of dosing
  Cmax
LNS8801 plasma exposure (t1/2) as a function of dose | During the first 23 days of dosing
  T1/2

CONTACTS AND LOCATIONS:
Overall Officials: Tina Garyantes, PhD, Study Director — Linnaeus Therapeutics, Inc.
Locations (10):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - The START Center for Cancer Care, San Antonio, Texas